CLINICAL TRIAL: NCT01167023
Title: A Double-Blind, Randomized, Multicenter Study of Prasugrel Compared to Placebo in Adult Patients With Sickle Cell Disease
Brief Title: Prasugrel Versus Placebo in Adult Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13806; H7T-MC-TAEK (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Results first posted 2012-05-03 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-04

CONDITIONS: Sickle Cell Anemia
Keywords: Sickle Cell Disease; Sickle Cell Anemia; Adult
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 7.5 mg Prasugrel (Experimental): Participants were to receive 7.5 milligrams (mg) of prasugrel orally, once daily if they weighed ≥60 kilograms (kg) and if pharmacodynamic (PD) measures indicated that the 5-mg prasugrel dose did not produce a steady-state PD response equivalent to inhibition of platelet activation (IPA) ≥25%. Because these criteria were not met, no participants received 7.5 mg of prasugrel.
  Interventions: Drug: Prasugrel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 5 mg Prasugrel (Experimental)
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Prasugrel — Administered orally, once daily for 30 days.
  Other Names: Efient; Effient; LY640315; CS747
  Arms: 5 mg Prasugrel; 7.5 mg Prasugrel
Drug: Placebo — Administered orally, once daily for 30 days.
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess the safety of Prasugrel in adult patients with sickle cell disease (SCD) by monitoring the rate and severity of hemorrhagic events requiring medical intervention compared to placebo for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Sickle Cell Disease (SCD).
* Are greater than or equal to 50 kilograms (kg) at time of screening.
* Are not currently being treated with an investigational drug (use of hydroxyurea, which is not an investigational drug, is permitted under this protocol if the patient has been on a stable dose for at least 30 days prior to randomization and has no signs of hematological toxicity at screening.
* Agree to use a reliable method of birth control during the study or are women not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause.

Exclusion Criteria:

* Acute painful crisis (requiring medical attention) within 30 days prior to screening.
* Have a concomitant medical illness (for example, terminal malignancy) that, in the opinion of the investigator, is associated with reduced survival over the expected treatment period (approximately 30 days).
* Severe hepatic dysfunction (cirrhosis, portal hypertension, or aspartate aminotransferase (AST) greater than or equal to 3x upper limit of normal [ULN]).
* Renal dysfunction requiring chronic dialysis.
* Contraindication for antiplatelet therapy.
* History of intolerance or allergy to approved thienopyridines.
* Have signs or symptoms of an infection.
* Hypertension (systolic blood pressure >180 millimeters of mercury (mm Hg) or diastolic blood pressure >110 mm Hg) at the time of screening or randomization.
* Hematocrit <18%.
* Any history of bleeding diathesis, bleeding requiring in-hospital treatment, or papillary necrosis.
* Active internal bleeding.
* History of spontaneous gastrointestinal (GI) bleeding requiring in-hospital treatment.
* Gross hematuria. Microhematuria, common in SCD patients, is not a contraindication.
* Platelet count <100,000 per cubic millimeter.
* Any history of intraocular hemorrhage.
* Prior history of transient ischemic attack (TIA), ischemic stroke, hemorrhagic stroke, or other intracranial hemorrhage.
* Known history of intracranial neoplasm, arteriovenous malformation, or aneurysm.
* Have clinical findings, in the judgment of the investigator, associated with an increased risk of bleeding.
* Have an international normalized ratio (INR) of greater than 1.5 at screening.
* Have had recent surgery (within 30 days prior to screening) or are scheduled to undergo surgery within the next 60 days.
* History of menorrhagia requiring medical intervention.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (14):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jenkintown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo orally, once daily for 30 days.
- 5 mg Prasugrel: Participants received 5 mg of prasugrel orally, once daily for 30 days.
Period: Overall Study
Arm/Group | 7.5 mg Prasugrel | Placebo | 5 mg Prasugrel
Started | 0 | 21 | 41
Received at Least 1 Dose of Study Drug | 0 | 19 | 41
Completed | 0 | 18 | 39
Not Completed | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Screen Failure | 0 | 1 | 0
Not completed — Sponsor Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 5 mg Prasugrel | Total
Number analyzed (Participants) | 21 | 41 | 62
Age Continuous [Mean (Standard Deviation); unit: years] | 31.52 (8.20) | 32.88 (8.60) | 32.42 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 21 | 30
  Male | 12 | 20 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 40 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 40 | 61
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 8 | 11
  United States | 18 | 33 | 51
Sickle-Cell Genotype [Number; unit: participants] — The number of participants for this baseline measure differs from the overall number of baseline participants because 1 participant from the 5-mg prasugrel arm did not have sickle cell disease (SCD), but possessed the thalassemia trait.
  participants
    Hb S ß+ thalassemia genotype | 2 | 4 | 6
    Hb S ß0 thalassemia genotype | 1 | 2 | 3
    Hb SC genotype | 5 | 10 | 15
    Hemoglobin SS (Hb SS) genotype | 13 | 24 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hemorrhagic Events Requiring Medical Intervention During the Treatment Duration
Description: A hemorrhagic event requiring medical intervention. Medical intervention was defined as any medical attention resulting in therapy or further investigation during the 30-day treatment duration.
Time Frame: Baseline through 30 days
Population: Safety population: All randomized participants who took at least 1 dose of study medication. Participants were analyzed according to the treatment they actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 5 mg Prasugrel
Number analyzed (Participants) | 19 | 41
percentage of participants | 0 | 0

2. Secondary Outcome: Percentage of Participants With Hemorrhagic Treatment-Emergent Adverse Events (TEAEs) During the Treatment Duration
Description: TEAEs were defined as AEs that occurred or worsened after receiving the study drug.
Time Frame: Baseline through 30 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 5 mg Prasugrel
Number analyzed (Participants) | 19 | 41
percentage of participants | 5.3 | 19.5

3. Secondary Outcome: Percentage of Days With Pain Related to Sickle Cell Disease (SCD) During the Treatment Duration
Description: Participants recorded the intensity of pain due to SCD each day in the daily pain diaries. A scale of 0 to 9 was used, with 0 indicating no pain, and 9 indicating unbearable pain. A response range of 1 to 9 indicated the participant experienced pain due to SCD, whereas a response of 0 indicated participant did not experience pain due to SCD. The percentage of days with pain (pain rate) was calculated as follows: Pain rate = 100*(Total number of days with pain/number of daily pain diaries completed). Number of daily pain diaries completed was number of nonmissing pain intensity responses.
Time Frame: Baseline through 30 days
Population: Intent to treat (ITT) population consisted of all randomized participants. Participants were analyzed according to the treatment they were randomized to. The analysis was performed in the ITT population who recorded pain intensity in at least 1 daily pain diary.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo | 5 mg Prasugrel
Number analyzed (Participants) | 18 | 40
percentage of days | 63.57 (41.80) | 39.04 (42.20)
Statistical Analysis 1: Comparison: Placebo vs 5 mg Prasugrel; Test type: Superiority or Other; p = 0.304, ANCOVA — Pain rate was analyzed using an analysis of covariance (ANCOVA) model, with baseline pain intensity, treatment group, and stratification variable sickle-cell genotype as explanatory variables; Least Squares Mean Difference = -11.26 — Least Squares (LS) Mean Difference is for 5 mg prasugrel minus placebo

4. Secondary Outcome: Percentage of Participants With Pain Events Related to Sickle Cell Disease (SCD) Requiring Medical Attention During the Treatment Duration
Description: Pain requiring medical attention was defined 2 ways: (1) if the participant attended an unplanned doctor's appointment or clinic visit, visited the emergency room, or was admitted to hospital due to sickle cell pain, or (2) if the participant experienced a vaso-occlusive crisis (VOC), acute chest syndrome, or hepatic sequestration at least once during the treatment period.
Time Frame: Baseline through 30 days
Population: Intent to treat (ITT) population consisted of all randomized participants. Participants were analyzed according to the treatment they were randomized to. The analysis was performed in the ITT population who completed at least 1 page of the daily pain diary or with pain endpoint case report form (CRF) data available.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 5 mg Prasugrel
Number analyzed (Participants) | 19 | 40
percentage of participants | 36.8 | 22.5

5. Secondary Outcome: Platelet Reactivity Index (PRI) Measured by Vasodilator-Associated Stimulated Phosphoprotein (VASP) at 30 Days
Description: PRI was calculated by VASP phosphorylation assay using flow cytometry. The PRI indicates the level of P2Y12 inhibition. A low PRI reflects strong inhibition of P2Y12, whereas a high PRI reflects weak/absent inhibition of P2Y12. The Least Squares (LS) Mean values were calculated from a mixed-effects model repeated measures (MMRM) analysis with baseline measurement, stratification variable sickle cell genotype, treatment, time, and time*treatment interaction as fixed effects, and participant as a random effect in the model.
Time Frame: 30 days
Population: All randomized participants who took at least 1 dose of study medication. Participants were analyzed according to the treatment they actually received. The analysis was performed in the safety population who had both baseline and 30-day PRI measurements and a non-missing genotype.
Measure: Least Squares Mean (Standard Error); unit: percentage of PRI
Arm/Group | Placebo | 5 mg Prasugrel
Number analyzed (Participants) | 14 | 30
percentage of PRI | 74.843 (4.993) | 50.792 (3.360)
Statistical Analysis 1: Comparison: Placebo vs 5 mg Prasugrel; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — A mixed-effects model repeated measures analysis with baseline measurement, stratification variable sickle cell genotype, treatment, time, and time*treatment interaction as fixed effects, and participant as a random effect in the model was used; Least Squares Mean Difference = -24.051 — Least Squares Mean Difference is for 5 mg prasugrel minus placebo

6. Secondary Outcome: Intensity of Pain Related to Sickle Cell Disease (SCD) During the Treatment Duration
Description: Participants recorded intensity of pain due to SCD each day in daily pain diaries using a pain scale. A scale of 0 to 9 was used, with 0=no pain and 9=unbearable pain. A response range of 1 to 9 indicated participant experienced pain due to SCD, whereas a response of 0 indicated participant did not experience pain due to SCD. Pain intensity was the average of a participant's pain ratings. Average pain intensity=(Sum of all nonmissing pain intensity responses/number of daily pain diaries completed). Number of daily pain diaries completed is number of nonmissing pain intensity responses.
Time Frame: Baseline through 30 days
Population: Intent to treat (ITT) population consisted of all randomized participants. Participants were analyzed according to the treatment they were randomized to. The analysis was performed in the ITT population who had recorded the pain intensity in at least 1 daily pain diary.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 5 mg Prasugrel
Number analyzed (Participants) | 18 | 40
units on a scale | 2.72 (2.33) | 1.56 (1.98)
Statistical Analysis 1: Comparison: Placebo vs 5 mg Prasugrel; Test type: Superiority or Other; p = 0.244, ANCOVA — Average pain intensity was analyzed using an analysis of covariance (ANCOVA) model, with baseline intensity, treatment group and stratification variable sickle-cell genotype as explanatory variables; Least Squares Mean Difference = -0.56 — Least Squares (LS) Mean Difference is for 5 mg prasugrel minus placebo

7. Secondary Outcome: P2Y12 Reaction Units (PRU) as Measured by Accumetrics VerifyNow® P2Y12 (VN P2Y12) at 30 Days
Description: PRU represents the rate and extent of adenosine (ADP)-stimulated platelet aggregation. The VN P2Y12 assay is a point-of-care device that measures platelet aggregation with single-use, disposable cartridges. A low PRU reflects stronger inhibition of P2Y12, whereas a high PRU reflects weaker inhibition of P2Y12. The Least Squares Mean values were calculated from a mixed-effects model repeated measures analysis with baseline measurement, stratification variable sickle cell genotype, treatment, time, and time*treatment interaction as fixed effects, and participant as a random effect in the model.
Time Frame: 30 days
Population: Safety population: All randomized participants who took at least 1 dose of study medication. Participants were analyzed according to the treatment they actually received. The analysis was performed in the safety population who had both baseline and 30-day PRU measurements and a non-missing genotype.
Measure: Least Squares Mean (Standard Error); unit: P2Y12 Reaction Units (PRU)
Arm/Group | Placebo | 5 mg Prasugrel
Number analyzed (Participants) | 18 | 35
P2Y12 Reaction Units (PRU) | 336.8 (16.8) | 208.5 (11.9)
Statistical Analysis 1: Comparison: Placebo vs 5 mg Prasugrel; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — A mixed-effects model repeated measures analysis with baseline measurement, stratification variable sickle cell genotype, treatment, time and time*treatment interaction as fixed effects, and participant as a random effect in the model; Least Squares Mean Difference = -128.3 — Least Squares (LS) Mean Difference is for 5 mg prasugrel minus placebo

ADVERSE EVENTS:
Arm/Group | Placebo | 5 mg Prasugrel
Serious Adverse Events (participants affected / at risk) | 4/19 | 8/41
Other Adverse Events (participants affected / at risk) | 16/19 | 33/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | 5 mg Prasugrel (N=41)
pain (General disorders) | 1 (1) | 0 (0)
pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
sickle cell anaemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 (1) | 2 (2)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)
osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
thrombosis (Vascular disorders) | 1 (1) | 0 (0)
vascular occlusion (Vascular disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | 5 mg Prasugrel (N=41)
fatigue (General disorders) | 2 (2) | 1 (1)
malaise (General disorders) | 1 (2) | 1 (2)
pain (General disorders) | 7 (7) | 11 (21)
anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 (0) | 3 (5)
ocular icterus (Eye disorders) | 1 (1) | 0 (0)
photophobia (Eye disorders) | 1 (1) | 0 (0)
visual impairment (Eye disorders) | 1 (1) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
gingival bleeding (Gastrointestinal disorders) | 1 (1) | 2 (4)
haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
jaundice (Hepatobiliary disorders) | 1 (1) | 2 (2)
drug hypersensitivity (Immune system disorders) | 1 (3) | 0 (0)
seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (1)
chorioretinal scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
sciatic nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
cardiac murmur (Investigations) | 1 (1) | 0 (0)
decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
dizziness (Nervous system disorders) | 1 (1) | 2 (2)
headache (Nervous system disorders) | 3 (3) | 5 (12)
priapism (Reproductive system and breast disorders) | 1 (1) | 0 (0)
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hot flush (Vascular disorders) | 1 (1) | 0 (0)
thrombosis (Vascular disorders) | 1 (1) | 0 (0)
vascular occlusion (Vascular disorders) | 4 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days